CLINICAL TRIAL: NCT05043818
Title: A Clinical Study on the Screening of Intestinal Biomarkers in IBD Patients With Depression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yanling Wei, Yanling Wei Deputy Chief Physician, Third Military Medical University
Other Study IDs: TMMU-DP-GI-IBD
Record Dates: First submitted 2021-08-09; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Ulcerative Colitis, Crohn's Disease，Anxiety ， Depression
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD patients with depression: IBD patients with depression
- IBD patients without depression: IBD patients without depression

INTERVENTIONS:
Other:  — This study is an observational study and does not involve intervention.When the patient comes to the hospital or on the first to the second day of admission, the subject will be given a full scale check once（Screening related scales for anxiety and depression symptoms (PHQ9, SDS, HADS, HAMA, HAMD), inflammatory bowel disease quality of life scale (IBDQ), modified Mayo score for patients with ulcerative colitis/ simplified CDAI score for patients with Crohn's disease , Stool characteristics, degree of abdominal pain, gastrointestinal symptom scale (GSRS), etc.）. The stool sample will be collected once and 16S rRNA sequencing.

SUMMARY:
Inflammatory bowel disease (IBD) seriously affects the quality of life of patients. During treatment, it is found that patients are often accompanied by a certain degree of psychological problems, such as depression, sensitivity, introversion, depression, and pessimistic disappointment. Among them, anxiety and depression are the most common. Through prospective observational research, statistics of the incidence of depression in inflammatory bowel disease in our hospital, comparison of the proportions of each subtype, screening of intestinal biomarkers in IBD patients with depression, and observation of inflammatory bowel disease with different The type and quantity of different intestinal flora in patients with severe depression, and the correlation between intestinal flora and depression.

DETAILED DESCRIPTION:
The subjects voluntarily participated in the study and signed an informed consent form. Follow the steps below:

1. When you come to the hospital or the first to second days of admission, collect general information: ID number, gender, age, height, weight, BMI, complete medical history including a) date of diagnosis, b) degree of disease, c) course of disease , D) previous surgery, e) previous hospitalization, f) comorbidities, g) current symptoms, h) extra-articular manifestations, i) endoscopic data, j) treatment drugs and other data.
2. Scale evaluation (see Annex 1 for details): Screening related scales for anxiety and depression symptoms (PHQ9, SDS, HADS, HAMA, HAMD), inflammatory bowel disease quality of life scale (IBDQ), ulcerative colitis Patient's modified Mayo score/Simplified questionnaire surveys for patients with Crohn's disease such as CDAI score, stool characteristics, abdominal pain degree, and Gastrointestinal Symptom Scale (GSRS);
3. Stool specimens were collected once during the visit to the hospital.
4. The time, frequency and precautions for patients to go to the hospital for examination and follow-up.

This trial is a prospective observational study. When the patient comes to the hospital or on the first to the second day of admission, the subject will be given a full set of scales to check once, and a stool sample will be collected during the treatment. Co., Ltd. performed 16S rRNA sequencing to analyze the results of the bacterial flora once. In this study, there is no need for patients to come to the hospital for follow-up follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of inflammatory bowel disease【diagnostic criteria reference: (2020)JSGE Evidence-based clinical practice guidelines: inflammatory bowel disease】
2. There is no restriction on men and women, aged 18-65 years old;
3. No complicated other serious diseases such as heart, brain, lung, liver, kidney, etc., no mental illness, and normal communication skills;
4. No antibiotics, Bifidobacterium, Bacillus subtilis and other probiotic preparations have been used within one month;
5. Sign the informed consent form and agree to participate in this research.

Exclusion Criteria:

1. Course of disease <6 months;
2. Unspecified inflammatory bowel disease.
3. Authors with bipolar disorder, persistent mood disorder, and mania;
4. Patients with malignant tumors;
5. Patients during pregnancy and lactation;
6. Combined with hypertension, diabetes, heart disease, stroke or severe chronic disease (infectious, genetic, metabolic, internal Secretory diseases);
7. Patients who cannot cooperate to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease diagnosed in the outpatient clinic or hospitalization of our hospital
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 score | 0 week
  Patient Health Questionnaire-9. The score varies from 0 to 27, higher scores suggest more severe the depression.Total score is the sum of 9 corresponding numbers:
  0-4 points: no depression; 5-9 points: mild depression; 10-14 points: moderate depression; 15-27 points: severe depression.

SECONDARY OUTCOMES:
SDS score | 0 week
  Self-rating Depression Scale. The score varies from 25 to 100. Higher scores suggest more severe depression.
HAMA-score | 0 week
  Hamilton Anxiety Scale.The total score is 0-56, among which, physical anxiety: 7-13 items; mental anxiety: 1-6 and 14 items.The higher the score, the greater the anxiety.
HAMD-score | 0 week
  Hamilton Depression Scale.The total score is 0-35 points: >35 points: severe depression; >20 points: mild or moderate depression; 8-20 may have depression; <8 points: no depression. The higher the score, the greater the anxiety.
HADS-score | 0 week
  Hospital Anxiety and Depression Scale.It consists of 14 (7 anxiety and 7 depression-related) scoring items, all ranging from 0-21. The higher the score, the more severe the anxiety and depression.
GSRS-score | 0 week
  Gastrointestinal Symptom Rating Scale. The score varies from 16 to 112. High scores suggest more severe Gastrointestinal pathology.
Simplified CDAI score | 0 week
  Simplified CDAI score for Crohn's disease: represents disease activity, <4 remission period 5~8 moderate activity> 9 heavy activity. The higher the score, the more severe the condition.
Modified Mayo score for UC | 0 week
  Modified Mayo score for ulcerative colitis: a total of 0-12 points, scores ≤ 2 points and no single sub-item score> 1 points to clinical remission, 3 to 5 points to mild activity, 6 to 10 points to moderate activity, 11 ~12 is divided into heavy activity.
IBD-QoL | 0 week
  Quality of Life Analysis Table for Patients with Inflammatory Bowel Disease: There are 32 questions in total. Each question has a different level of answer from 1 to 7, 1 generation The table has the heaviest degree, and 7 represents the least degree.

OTHER OUTCOMES:
Intestinal flora | 0 week
  Use metagenomics technology to detect intestinal flora.

CONTACTS AND LOCATIONS:
Overall Officials: Yanling Wei, MD, Principal Investigator — Army Medical Center of PLA
Locations (1):
- Department of Gastroenterology, Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China